CLINICAL TRIAL: NCT06368401
Title: Transcatheter Tricuspid Repair Utilizing the Versa Vascular Repair System
Brief Title: A First in Human Study for the Versa Device for Tricuspid Regurgitation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Versa Vascular, Inc (Industry)
Collaborators: Cardiovascular Research Foundation, New York (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: TP_01428
Record Dates: First submitted 2024-04-07; First posted 2024-04-16 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Tricuspid Regurgitation
MeSH Terms: conditions — Tricuspid Valve Insufficiency

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Implant (Experimental): Participants who pass all screening criteria will undergo a percutaneous procedure for the implantation of a permanent tricuspid repair device. Participants will be followed for 1 year to evaluate the safety and feasibility of the Versa System procedure and the Versa Tricuspid Repair Implant.
  Interventions: Device: Versa Implant

INTERVENTIONS:
Device: Versa Implant — The Versa Vascular Implant and Delivery System consists of a percutaneously delivered, permanent right-atrial implant and the delivery catheter that is used to first position the implant over the native valve orifice and to then place the implant.

SUMMARY:
This study is prospective, non-randomized, single-arm,first in human study to evaluate the safety and feasibility of the Versa Vascular System for intervention in adults with severe tricuspid regurgitation who are not surgical candidates.

ELIGIBILITY:
Inclusion Criteria:

* Tricuspid regurgitation (TR) associated symptoms despite optimal medical treatment.
* TR ≥ 3 as determined by the assessment of a transthoracic echocardiogram or transesophageal echocardiogram.
* The local multi-disciplinary heart team agrees that the participant is a poor candidate for surgery.
* Age ≥ 18 years at the time of consent.
* Ability and willingness to provide written informed consent prior to any study related procedure(s).

Exclusion Criteria:

* Severe pulmonary hypertension.
* Severe uncontrolled hypertension Systolic Blood Pressure (SBP) ≥ 180 mmHg and/or Diastolic Blood Pressure (DBP) ≥ 110 mmHg.
* Any condition that would interfere with the Versa procedure, such as prior tricuspid valve repair or tricuspid valve leaflet anatomy which may preclude successful device implantation, pacemaker or Implantable Cardioverter Defibrillator (ICD) leads that would prevent appropriate placement or visualization of Versa implant, Ebstein Anomaly (normal annulus position, but valve leaflets attached to walls and septum of the right ventricle), tricuspid valve anatomy non-evaluable by echocardiography.
* Known allergy to antiplatelet therapy, heparin, or to device materials.
* Femoral venous mass or thrombus or vegetation.
* Tricuspid valve anatomy not compatible with the Versa implant
* Undergone any heart valve surgery within prior 60 days.
* Tricuspid valve stenosis - Defined as a tricuspid valve orifice of ≤ 4.0 cm2.
* Severe mitral regurgitation.
* Left Ventricular Ejection Fraction (LVEF) ≤ 20%
* Active endocarditis, other ongoing infection requiring antibiotic therapy.
* Myocardial infarction or percutaneous coronary intervention within prior 30 days.
* Cardiogenic shock or the need for inotropic support or hemodynamic support device (e.g., intra-aortic balloon pump).
* Cerebrovascular Accident (CVA) within prior 30 days
* Active gastrointestinal (GI) bleeding
* Life expectancy of less than 12 months independent of tricuspid valvular disease.
* Subject currently participating in another clinical study (not yet completed primary endpoint).
* Pregnant or nursing subjects or those who plan pregnancy during the study.
* The presence of anatomic or comorbid conditions, or other medical, social, or psychological conditions that, in the eye of the investigator, limits the subject's ability to participate in the clinical investigation or comply with follow-up requirements.
* Absence of appropriate venous access.
* Unwillingness to complete the required follow-up visits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-08-05 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-10-02 (Estimated)

PRIMARY OUTCOMES:
Acute Procedural Success | Immediately after the procedure
  Successful in Versa Vascular Device implantation, and residual TR grade equivalent to a reduction of at least 1 grade of TR when compared to TR evaluated prior to implantation of the Versa Vascular Device.
Incidence of major adverse events (MAE) | (up to 7 days) from date of procedure to date of patient discharge from hospital
  Freedom from procedure and/or device related Major Adverse Events (MAE). MAE are defined as all-cause mortality, reoperation, or reintervention for tricuspid regurgitation prior to hospital discharge.

SECONDARY OUTCOMES:
Tricuspid Regurgitation Severity Change | 90 days
  Percentage of patients with tricuspid regurgitation reduced by at least one grade. Echocardiographic analysis of Tricuspid regurgitation at 90 days. TR grade at day 90 will be compared against TR grade at the time of implantation.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Webster, MD, Principal Investigator — Auckland City Hospital
Locations (2):
- Pontificia Universidad Católica, Santiago, Chile
- Auckland City Hospital, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No